CLINICAL TRIAL: NCT02500368
Title: A Dispensing Clinical Trial of a Study Test Silicone Hydrogel Lens Against Control Lens Over 1 Week
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CV-15-36
Record Dates: First submitted 2015-07-14; First posted 2015-07-16 (Estimated); Results first posted 2017-02-17 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- silicone hydrogel lens (test) (Experimental): Participants were randomized to wear silicone hydrogel lens (test) for 1 week during the cross over study.
  Interventions: Device: silicone hydrogel lens (test)
- enfilcon A lens (control) (Active Comparator): Participants were randomized to wear enfilcon A lens (control) for 1 week during the cross over study.
  Interventions: Device: enfilcon A lens (control)

INTERVENTIONS:
Device: silicone hydrogel lens (test) — contact lens
  Arms: silicone hydrogel lens (test)
Device: enfilcon A lens (control) — contact lens
  Arms: enfilcon A lens (control)

SUMMARY:
This is a 1-week dispensing, double-masked, randomized, bilateral study comparing the test lens against the control lens.

DETAILED DESCRIPTION:
The order of lens wear (test lens first, control lens second or control lens first, test lens second) will be selected according to a randomization table.

Both test and control lenses will be used in a daily wear modality for 1 week. It is anticipated that this study will involve following visits: Baseline (screening and dispense of 1st study pair of lenses, visit combined), 1-week visit (follow-up of the 1st study pair of lenses and dispense the 2nd study pair of lenses) and 2-week visit (1 week follow-up of the 2nd study pair of lenses).

ELIGIBILITY:
Inclusion criteria:

-A person is eligible for inclusion in the study if he/she:

* Is at least 17 years of age and has full legal capacity to volunteer
* Has read and understood the information consent letter
* Is willing and able to follow instructions and maintain the appointment schedule
* Is correctable to a visual acuity of 20/30 or better (in each eye) with their habitual correction and the assigned study lenses
* Is an adapted soft contact lens wearer (For the purpose of this study: Current lens wear at least 3 days per week, 8 hours each day.)

Exclusion Criteria:

-A person will be excluded from the study if he/she:

* Is participating in any concurrent clinical or research study
* Has any known active* ocular disease and/or infection
* Has a systemic condition that in the opinion of the investigator may affect a study outcome variable**
* Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable
* Has known sensitivity to the diagnostic pharmaceuticals to be used in the study
* Is pregnant, lactating or planning a pregnancy at the time of enrolment (by verbal confirmation at the screening visit).
* Is aphakic
* Has undergone corneal refractive surgery.

For the purposes of this study, active* ocular disease is defined as infection or inflammation which requires therapeutic treatment. Mild (i.e. not considered clinically relevant) lid abnormalities (blepharitis, meibomian gland dysfunction, papillae), corneal and conjunctival staining and dry eye are not considered active ocular disease. Neovascularization and corneal scars are the result of previous hypoxia, infection or inflammation and are therefore not active. Participants will be excluded with significant slit lamp findings (e.g. infiltrates or other slit lamp findings Grade 3 or above: corneal edema, tarsal abnormalities, and conjunctival injection) or active ocular disease (e.g. glaucoma, history of recurrent corneal erosions, and intraocular infection or inflammation of an allergic, bacterial, or viral etiology)

For the purposes of this study, participants will be excluded**, if currently taking medication, such as oral antihistamines, antihistamine eye drops, oral and ophthalmic beta-adrenergic blockers (e.g. Propanolol, Timolol), anticholinergics, oral steroids and any prescribed or over-the-counter eye medication, except artificial tears or eye lubricants

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-07; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD FCO, Principal Investigator — Center for Contact Lens Research, University of Waterloo
Locations (1):
- Center for Contact Lens Research, University of Waterloo, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant discontinued from the study as a screen failure before lens randomization.
Groups:
- Silicone Hydrogel Lens (Test), Then Enfilcon A Lens (Control): Participants were randomized to wear silicone hydrogel lens (test) for 1 week, then cross over to the enfilcon A lens (control).
  silicone hydrogel lens (test): contact lens
  enfilcon A lens (control): contact lens
- Enfilcon A Lens (Control), Then Silicone Hydrogel Lens (Test): Participants were randomized to wear enfilcon A lens (control) for 1 week, then cross over to the silicone hydrogel lens (test).
  enfilcon A lens (control): contact lens
  silicone hydrogel lens (test): contact lens
Period: First Intervention (1 Week)
Arm/Group | Silicone Hydrogel Lens (Test), Then Enfilcon A Lens (Control) | Enfilcon A Lens (Control), Then Silicone Hydrogel Lens (Test)
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: Second Intervention (1 Week)
Arm/Group | Silicone Hydrogel Lens (Test), Then Enfilcon A Lens (Control) | Enfilcon A Lens (Control), Then Silicone Hydrogel Lens (Test)
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Baseline Characteristics: Participants were randomized to wear silicone hydrogel lens (test) or enfilcon A lens (control) for 1 week during the cross over study.
Arm/Group | Overall Baseline Characteristics
Number analyzed (Participants) | 41
Age, Continuous [Median (Full Range); unit: years] | 24 [19 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Comfort
Description: Subjective ratings scale (0-100) assessed: 0=Cannot be worn, causes pain, 20=Frequently irritating, 40=Occasionally irritating, 60=Occasionally noticable but not irritating, 80=Rarely noticeable, 100=Cannot be felt ever. Time points for comfort: lens dispense at baseline, lens insertion at 1 week, and overall at 1 week.
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Silicone Hydrogel Lens (Test) | Enfilcon A Lens (Control)
Number analyzed (Participants) | 40 | 40
units on a scale
  Lens dispense at baseline | 90 (11) | 91 (10)
  Lens insertion at 1 week | 92 (9) | 90 (14)
  Overall comfort at 1 week | 79 (15) | 81 (13)

2. Primary Outcome: Dryness
Description: Subjective ratings scale (0-100): 0=Cannot be worn, extremely dry, 20=Frequently Irritating, 40=Occasionally irritating, 60=Occasionally noticeable but not irritating, 80=Rarely noticeable, 100=No dryness experienced at any time. Time points for dryness: lens dispense at baseline, lens insertion at 1 week, and overall at 1 week.
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Silicone Hydrogel Lens (Test) | Enfilcon A Lens (Control)
Number analyzed (Participants) | 40 | 40
units on a scale
  Lens dispense at baseline | 94 (10) | 94 (10)
  Lens insertion at 1 week | 94 (8) | 92 (12)
  Overall dryness at 1 week | 75 (19) | 78 (16)

3. Secondary Outcome: Lens Wettability
Description: Grading scale 0-4, 0.25 steps, 0=excellent; 4=severely reduced.
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Silicone Hydrogel Lens (Test) | Enfilcon A Lens (Control)
Number analyzed (Participants) | 40 | 40
units on a scale
  Baseline | 1.09 (0.60) | 1.18 (0.87)
  1 week | 1.17 (0.76) | 1.38 (0.79)

4. Secondary Outcome: Surface Appearance
Description: Grade ratings category (smooth, grainy, or other)
Time Frame: Baseline
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Silicone Hydrogel Lens (Test) | Enfilcon A Lens (Control)
Number analyzed (Participants) | 40 | 40
Number analyzed (Eyes) | 80 | 80
Eyes
  Smooth | 76 | 70
  Grainy | 3 | 4
  Other | 1 | 6

5. Secondary Outcome: Surface Appearance
Description: Grade ratings category (smooth, grainy, or other)
Time Frame: 1 week
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Silicone Hydrogel Lens (Test) | Enfilcon A Lens (Control)
Number analyzed (Participants) | 40 | 40
Number analyzed (Eyes) | 80 | 80
Eyes
  Smooth | 77 | 72
  Grainy | 1 | 4
  Other | 2 | 4

6. Secondary Outcome: High Contrast Acuity at High Room Illumination
Description: Logarithm of the Minimum Angle or Resolution (LogMAR) Chart
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Silicone Hydrogel Lens (Test) | Enfilcon A Lens (Control)
Number analyzed (Participants) | 40 | 40
LogMAR
  Baseline | -0.10 (0.06) | -0.09 (0.04)
  1 week | -0.10 (0.05) | -0.08 (0.06)

7. Secondary Outcome: Lens Deposition
Description: Lens Deposits Scale 0-4, 0.25 steps. 0=excellent; 4=severely reduced
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Silicone Hydrogel Lens (Test) | Enfilcon A Lens (Control)
Number analyzed (Participants) | 40 | 40
units on a scale
  Baseline | 0.06 (0.13) | 0.12 (0.21)
  1 week | 0.28 (0.32) | 0.38 (0.48)

8. Secondary Outcome: Lens Problems
Description: Lenses were evaluated for defects, scratches, fibers, blue specks, and other findings.
Time Frame: Baseline and 1 week
Measure: Number; unit: Lenses
Units Other Than Participants: Lenses
Arm/Group | Silicone Hydrogel Lens (Test) | Enfilcon A Lens (Control)
Number analyzed (Participants) | 40 | 40
Number analyzed (Lenses) | 80 | 80
Lenses
  Baseline, Blue specs | 0 | 2
  Baseline, Fibers | 0 | 1
  Baseline, Nick | 0 | 1
  1 week, Blue specs | 0 | 2
  1 week, Nick | 0 | 1
  1 week, Particles | 0 | 3

9. Secondary Outcome: Lens Centration
Description: Lens centration was evaluated by the conjunctival overlap to determine whether lens was slightly or excessively decentered.
  (mm, 0.1 steps) N - Nasal, T - Temporal, S - Superior, I - Interior, N/S - Nasal/Superior, N/I - Nasal/Interior, T/S - Temporal/Superior T/I - Temporal/Interior
Time Frame: Baseline
Measure: Number; unit: eyes
Units Other Than Participants: Eyes
Arm/Group | Silicone Hydrogel Lens (Test) | Enfilcon A Lens (Control)
Number analyzed (Participants) | 40 | 40
Number analyzed (Eyes) | 80 | 80
eyes
  No decentration | 46 | 32
  N | 4 | 3
  T | 16 | 16
  S | 6 | 6
  I | 4 | 11
  N/S | 0 | 0
  N/I | 0 | 2
  T/S | 2 | 6
  T/I | 2 | 4

10. Secondary Outcome: Lens Centration
Description: as for outcome 9
Time Frame: 1 week
Measure: Number; unit: eyes
Units Other Than Participants: Eyes
Arm/Group | Silicone Hydrogel Lens (Test) | Enfilcon A Lens (Control)
Number analyzed (Participants) | 40 | 40
Number analyzed (Eyes) | 80 | 80
eyes
  No decentration | 43 | 51
  N | 1 | 1
  T | 12 | 6
  S | 8 | 4
  I | 10 | 9
  N/S | 1 | 0
  N/I | 1 | 0
  T/S | 3 | 2
  T/I | 1 | 7

11. Secondary Outcome: Post-blink Movement
Description: Post-blink movement evaluated by estimating the distance the lens was moving immediately after a blink. Primary Gaze: (mm, 0.1 steps)
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: mm steps
Arm/Group | Silicone Hydrogel Lens (Test) | Enfilcon A Lens (Control)
Number analyzed (Participants) | 40 | 40
mm steps
  Baseline | 0.26 (0.16) | 0.25 (0.10)
  1 week | 0.24 (0.10) | 0.27 (0.13)

12. Secondary Outcome: Lens Tightness
Description: Lens tightness Scale 0%-100%, 0%=extremely loose fit, 50%=optimal push resistance and smooth return, 100%=no movement.
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: percentage of tightness
Arm/Group | Silicone Hydrogel Lens (Test) | Enfilcon A Lens (Control)
Number analyzed (Participants) | 40 | 40
percentage of tightness
  Baseline | 50.9 (7.8) | 48.1 (6.3)
  1 week | 48.8 (9.1) | 47.9 (6.4)

13. Secondary Outcome: Visual Quality
Description: Subjective ratings scale (0-100): 0=Extremely poor vision all of the time; cannot function, 20=Frequently annoying vision problems, 40=Occasionally annoying vision problems, 60=Occasionally noticeable but not annoying vision problems, 80=Rarely noticeable vision problems, 100=Excellent vision all of the time. Different time points were taken for vision quality: lens dispense at baseline, lens insertion at 1 week, and overall at 1 week.
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Silicone Hydrogel Lens (Test) | Enfilcon A Lens (Control)
Number analyzed (Participants) | 40 | 40
units on a scale
  Lens dispense at baseline | 94 (7) | 93 (9)
  Lens insertion at 1 week | 95 (7) | 94 (9)
  Overall vision quality at 1 week | 88 (12) | 88 (13)

14. Secondary Outcome: Ease of Lens Insertion
Description: Subjective ratings scale (0-100): 0=Could not place lens on eye, 20=Frequently takes multiple attempts to place on eye; often unsuccessful, 40=Frequently takes multiple attempts to place on eye, 60=Occasionally takes a few attempts to place on eye, 80=Rarely difficult to place on eye, 100=Always easy to place lens on eye
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Silicone Hydrogel Lens (Test) | Enfilcon A Lens (Control)
Number analyzed (Participants) | 40 | 40
units on a scale
  Baseline | 97 (5) | 92 (10)
  1 week | 91 (9) | 90 (10)

15. Secondary Outcome: Ease of Lens Removal
Description: Subjective ratings scale (0-100): 0=Could not remove lens from eye, 20=Frequently takes multiple attempts to remove from eye; often unsuccessful, 40=Frequently takes multiple attempts to remove from eye, 60=Occasionally takes a few attempts to remove from eye, 80=Rarely difficult to remove from eye, 100=Always easy to remove lens from eye.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Silicone Hydrogel Lens (Test) | Enfilcon A Lens (Control)
Number analyzed (Participants) | 40 | 40
units on a scale | 86 (15) | 90 (12)

16. Secondary Outcome: Overall Lens Fit
Description: Overall Lens Fit Scale 0-4, 0.25 steps 0=Very poor (lens should not be worn at all);
  1. Poor (lens could be worn with supervision only);
  2. Fair (would prefer to refit, but clinically acceptable);
  3. Good (fit could be slightly improved);
  4. Very good (optimal)
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Silicone Hydrogel Lens (Test) | Enfilcon A Lens (Control)
Number analyzed (Participants) | 40 | 40
units on a scale
  Baseline | 3.35 (0.42) | 3.33 (0.36)
  1 week | 3.36 (0.41) | 3.38 (0.48)

17. Secondary Outcome: Bulbar Hyperemia
Description: Bulbar hyperemia assessed using scale 0-4, 0.5 steps, 0=No hyperemia, 4=Severe hyperemia.
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Silicone Hydrogel Lens (Test) | Enfilcon A Lens (Control)
Number analyzed (Participants) | 40 | 40
units on a scale
  Baseline | 1.96 (0.50) | 1.96 (0.50)
  1 week | 1.87 (0.44) | 1.95 (0.41)

18. Secondary Outcome: Limbal Hyperemia
Description: Limbal hyperemia assessed using scale 0-4, 0.5 steps, 0=No hyperemia, 4=Severe hyperemia.
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Silicone Hydrogel Lens (Test) | Enfilcon A Lens (Control)
Number analyzed (Participants) | 40 | 40
units on a scale
  Baseline | 1.76 (0.51) | 1.76 (0.51)
  1 week | 1.68 (0.42) | 1.71 (0.37)

19. Secondary Outcome: Corneal Dehydration Staining
Description: Corneal Staining: Dehydration Staining: Yes/No
Time Frame: 1 week
Measure: Number; unit: participants
Arm/Group | Silicone Hydrogel Lens (Test) | Enfilcon A Lens (Control)
Number analyzed (Participants) | 40 | 40
participants
  Both eyes | 3 | 1
  One eye | 2 | 2

20. Secondary Outcome: Corneal Staining (Extent)
Description: Corneal staining extent, grade as % of each zone:
  C - Central, N - Nasal, T - Temporal, S - Superior, I - Interior
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: percentage of cornea
Arm/Group | Silicone Hydrogel Lens (Test) | Enfilcon A Lens (Control)
Number analyzed (Participants) | 40 | 40
percentage of cornea
  Central - baseline | 1.21 (4.97) | 1.21 (4.97)
  Central - 1 week | 0.64 (1.73) | 0.75 (4.97)
  Nasal - baseline | 4.76 (9.10) | 4.76 (9.10)
  Nasal - 1 week | 2.20 (6.68) | 1.43 (4.79)
  Temporal - baseline | 2.04 (5.47) | 2.04 (5.47)
  Temporal - 1 week | 1.38 (4.05) | 1.04 (2.92)
  Superior - baseline | 2.15 (7.21) | 2.15 (7.21)
  Superior - 1 week | 1.75 (4.42) | 0.69 (2.07)
  Inferior - baseline | 5.88 (10.85) | 5.88 (10.85)
  Inferior - 1 week | 6.48 (11.52) | 5.01 (9.23)

21. Secondary Outcome: Conjunctival Indentation
Description: Conjunctival Indentation 5 locations (central, nasal, temporal, superior, inferior): Scale 0-4, 0.5 steps; 0=None, 1=Trace, 2=Mild, 3=Moderate, 4=Severe
Time Frame: Baseline and 1 week.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Silicone Hydrogel Lens (Test) | Enfilcon A Lens (Control)
Number analyzed (Participants) | 40 | 40
units on a scale
  Nasal - baseline | 0.01 (0.11) | 0.01 (0.11)
  Nasal - 1 week | 0.36 (0.64) | 0.01 (0.06)
  Temporal - baseline | 0.00 (0.00) | 0.00 (0.00)
  Temporal - 1 week | 0.39 (0.68) | 0.02 (0.10)
  Superior - baseline | 0.00 (0.00) | 0.00 (0.00)
  Superior - 1 week | 0.21 (0.49) | 0.02 (0.10)
  Inferior - baseline | 0.00 (0.00) | 0.00 (0.00)
  Inferior - 1 week | 0.34 (0.67) | 0.03 (0.15)

22. Secondary Outcome: Conjunctival Staining
Description: Conjunctival Staining 5 locations (central, nasal, temporal, superior, inferior): Scale 0-4; 0.5 steps, 0=None,1=Minimal diffuse punctuate, 2=Coalescent punctuate, 3=Confluent, 4=Deep confluent
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Silicone Hydrogel Lens (Test) | Enfilcon A Lens (Control)
Number analyzed (Participants) | 40 | 40
units on a scale
  Nasal - baseline | 0.48 (0.45) | 0.48 (0.45)
  Nasal - 1 week | 0.67 (0.58) | 0.46 (0.40)
  Temporal - baseline | 0.47 (0.49) | 0.47 (0.49)
  Temporal - 1 week | 0.72 (0.63) | 0.55 (0.43)
  Superior - baseline | 0.12 (0.29) | 0.12 (0.29)
  Superior - 1 week | 0.25 (0.38) | 0.14 (0.26)
  Inferior - baseline | 0.23 (0.38) | 0.23 (0.38)
  Inferior - 1 week | 0.49 (0.52) | 0.32 (0.37)

ADVERSE EVENTS:
Time Frame: From dispense up to one week for each study lenses
Arm/Group | Silicone Hydrogel Lens (Test) | Enfilcon A Lens (Control)
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other